CLINICAL TRIAL: NCT06645808
Title: The Safety, Tolerability and Biodistribution of a Single Intravenous Administration of Two Zirconium-89 Labelled Vartumabs (F8scFV or C9scFv) in Patients With Solid Tumors - a Phase 0, Open Label, PET/CT Molecular Imaging Basket Trial
Brief Title: PET-imaging of Two Vartumabs in Patients With Solid Tumors
Acronym: VARTUTRACE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Var2 Pharmaceuticals (Industry)
Collaborators: TRACER Europe BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VAR2-2024-CS01; 2024-513827-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-28; First posted 2024-10-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Colon Carcinoma; Rectal Carcinoma; Osteosarcoma; Chondrosarcoma; Lung Carcinoma; Head and Neck Squamous Cell Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Pancreas Carcinoma; Bladder Carcinoma; Glioblastoma; Soft Tissue Sarcoma (STS); Breast Cancer
Keywords: Basket-trial; Oncology; Solid tumors
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Osteosarcoma; Chondrosarcoma; Lung Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Glioblastoma; Sarcoma; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Initially, three patients per compound (89Zr-C9scFv and 89Zr-F8scFv) will be included according to alternating inclusion or patient availability (n=6). Subsequently, an interim analysis will be conducted to determine the optimal radiation dose and optimal scanning day for each radiolabeled antibody fragment.
  After the interim analysis, cohorts will be expanded with additional solid tumor indications and will include 13 more subjects per compound (n=26), resulting in 32 subjects overall. This basket trial aims to include at least one patient per indication.
  For expansion cohort subjects, IMP-administration will occur on day 1, with one PET/CT scan performed on the most optimal day (this was determined to be day 4). Optionally, patients can receive an additional day 6 scan to gain more insight into tumor retention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 89Zr-F8scFv (Experimental): The first 3 patients of this arm will receive a single i.v. microdose (1 mg) administration of 89Zr-F8scFv 15 MBq, followed by three whole-body PET/CT scans on day 1, 2 and 4. After the first three patients, an interim analysis will be conducted to determine the optimal scanning time point and radiation dose.
  The following 13 patients will receive a single i.v. microdose administration of 89Zr-F8scFv between 15 - 30 MBq, followed by one whole-body PET/CT scan on the optimal scanning day (day 1-7). Each subject will have a follow-up visit approximately 28 days after IMP administration.
  Interventions: Biological: 89Zr-DFO-N-Suc-F8scFv; Radiation: PET/CT scan
- 89Zr-C9scFv (Experimental): The first 3 patients of this arm will receive a single i.v. microdose (1 mg) administration of 89Zr-C9scFv 15 MBq, followed by three whole-body PET/CT scans on day 1, 2 and 4. After the first three patients, an interim analysis will be conducted to determine the optimal scanning time point and radiation dose.
  The following 13 patients will receive a single i.v. microdose administration of 89Zr-C9scFv between 15 - 30 MBq, followed by one whole-body PET/CT scan on the optimal scanning day (day 1-7). Each subject will have a follow-up visit approximately 28 days after IMP administration.
  Interventions: Biological: 89Zr-DFO-N-Suc-C9scFv; Radiation: PET/CT scan

INTERVENTIONS:
Biological: 89Zr-DFO-N-Suc-F8scFv — 89-Zirconium labeled short-chain variable fragment F8 targeting oncofetal CS.
  Arms: 89Zr-F8scFv
Biological: 89Zr-DFO-N-Suc-C9scFv — 89-Zirconium labeled short-chain variable fragment C9 targeting oncofetal CS.
  Arms: 89Zr-C9scFv
Radiation: PET/CT scan — IMP administration will be followed by PET/CT scans on day 1, 2 and 4.

SUMMARY:
VARTUTRACE is a first-in-human PET/CT molecular imaging study in patients with solid tumors. This study will investigate the biodistribution and pharmacology of two antibody fragments binding oncofetal Chondroitin Sulfate (CS).

Oncofetal CS are tumor-specific carbohydrate motifs present in proteoglycans and identified by VAR2 Pharmaceuticals as expressed during fetal development. Oncofetal CS reappears in the vast majority of cancers while remaining largely absent from normal tissues.

VAR2 Pharmaceuticals recently developed antibodies specific for oncofetal CS. VARTUTRACE uses two of these as radiolabeled antibody fragments to study biodistribution, tumor accumulation, pharmacodynamics and clearance pathways in a diverse patient population.

DETAILED DESCRIPTION:
VARTUTRACE aims to investigate the biodistribution and pharmacology in patients with solid tumors of two antibody fragments specific for oncofetal CS.

VAR2 Pharmaceuticals has identified and characterized oncofetal CS as a group of tumor-specific carbohydrate motifs that appear in placental tissue during fetal development and in most cancers while remaining largely absent from healthy tissue. VAR2 Pharmaceuticals recently developed a panel of antibodies specific for oncofetal CS and characterized their tumor specificity, therapeutic, and safety in pre-clinical models under various formats.

VARTUTRACE is a Phase 0 microdosing study of a single administration of <30 nmol of one of the two most promising antibody fragments identified by VAR2 Pharmaceuticals - C9 and F8. Both antibody fragments will be used as short chain variable fragments (scFvs) labelled with the radioisotope Zirconium-89 (89Zr) and are therefore respectively named 89Zr-C9scFv or 89Zr-F8scFv. As it remains unclear from the pre-clinical in vitro and in vivo data which of the two will have the most optimal tumor targeting properties in patients with solid tumors, both scFvs will be evaluated.

The biodistribution, pharmacokinetics, pharmacodynamics, and clearance of two of these antibody fragments is planned to be studied in up to 32 patients with various cancers (i.e. a basket-trial).

ELIGIBILITY:
General Inclusion Criteria:

1. Willing to adhere to the prohibitions and restrictions specified in this protocol.
2. Capable of giving signed informed consent (voluntarily), indicating that the patient understands the purpose and procedures required for the study and is willing to comply with the requirements and restrictions listed in the informed consent form and in this protocol.
3. Patients aged ≥ 18 years at moment of signing informed consent form.
4. Life expectancy of > 12 weeks.
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
6. BMI ≥ 18.0 and ≤ 35.0 kg/m2 and weight at least 50 kg and no more than 120 kg at screening.
7. Overtly healthy based on medical history, physical findings, vital signs, ECG at the time of screening, as judged by the Investigator. Note: one retest of vital functions and ECG is allowed within the screening window.
8. Adequate liver- and kidney function, defined by the following laboratory results obtained during screening visit:

   * AST, ALT, and alkaline phosphatase ≤ 2.5x the upper limit of normal (ULN) as determined by the UMCG laboratory reference values.
   * Serum bilirubin ≤ 2.0x ULN as determined by the UMCG laboratory reference values. Patients with known Gilbert disease who have serum bilirubin level ≤ 3x ULN may be enrolled.
   * INR or APTT ≤ 1.5x ULN as determined by the UMCG laboratory reference values. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   * eGFR (based on plasma-creatinine) = >30 mL/min.
   * Serum albumin >35 g/L.
9. No other clinically significant laboratory abnormalities as determined by the investigator. Note: one retest of lab tests is allowed within the screening window.
10. Female patients should be at least 1 year post-menopausal (amenorrhea >12 months and/or follicle-stimulating hormone >30 mIU/mL) at screening or surgically sterile (bilateral oophorectomy, hysterectomy, or tubal ligation).
11. Male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control, and must not donate sperm, until 3 months after administration of 89Zr-DFO-N-Suc-scFv (F8 or C9).

Medical inclusion Criteria:

Colon Carcinoma:

1. Patients diagnosed with colon carcinoma stage I-IV, according to the 8th edition of the TNM-classification.
2. Histologically confirmed diagnosis of colon carcinoma.
3. Neo-adjuvant treatment according to the standard of care.

Rectal Carcinoma:

1. Patients diagnosed with rectal carcinoma stage I-IV, according to the 8th edition of the TNM-classification.
2. Histologically confirmed diagnosis of rectal carcinoma.
3. Neo-adjuvant treatment according to the standard of care.

Bone- and soft-tissue sarcoma

1. Patients diagnosed with a bone- or soft-tissue sarcoma stage I-IV, according to AJCC staging for Sarcoma.
2. Histologically confirmed diagnosis of sarcoma.
3. Neo-adjuvant treatment according to the standard of care.

Breast carcinoma

1. Patients diagnosed with breast carcinoma stage I-IV, according to the 8th edition of the TNM-classification.
2. Histologically confirmed diagnosis of breast carcinoma.
3. Neo-adjuvant treatment according to the standard of care.

Lung Carcinoma:

1. Anticipated diagnosis of Non-Small Cell Lung Carcinoma (NSCLC) stage I-IV, according to the 8th edition of the TNM-classification, based on imaging modalities such as (PET)/CT or based on cytology.
2. Neo-adjuvant treatment according to the standard of care.

Head and Neck Squamous Cell carcinoma (HNSCC):

1. Patients diagnosed with HNSCC of the oral cavity, oropharynx, nasal cavity, nasopharynx, hypopharynx and larynx.
2. Histologically confirmed diagnosis of HNSCC.
3. Neo-adjuvant treatment according to the standard of care.

Oesophageal and gastric carcinoma:

1. Patients diagnosed with oesophagus carcinoma stage I-IV according to the 7th edition of the TNM-classification.
2. Patients diagnosed with gastric carcinoma stage I-IV according to the 7th edition of the TNM-classification.
3. Histologically confirmed diagnosis of oesophageal- or gastric carcinoma.
4. Neo-adjuvant treatment according to the standard of care.

Pancreas carcinoma:

1. Anticipated diagnosis of pancreas carcinoma stage I-IV according to the 8th edition of the TNM-classification, based on imaging modalities such as (PET)/CT or based on cytology.
2. Histologically or cytologically confirmed diagnosis of pancreas carcinoma.
3. Neo-adjuvant treatment according to the standard of care.

Bladder carcinoma:

1. Patients diagnosed with invasive bladder carcinoma stage I-IV according to the 7th edition of the TNM-classification.
2. Histologically confirmed diagnosis of bladder carcinoma.
3. Neo-adjuvant treatment according to the standard of care.

Glioblastoma:

1. Anticipated diagnosis of a high-grade glioma (glioblastoma, grade 4 according to the WHO classification) based on imaging modalities such as MRI and/or CT or a biopsy.
2. Karnofsky performance status of at least 70%.
3. Neo-adjuvant treatment according to the standard of care.

General Exclusion Criteria:

1. Behavioral or cognitive impairment or psychiatric disease that, in the investigator's opinion, affects the patient's ability to understand and cooperate with the study protocol.
2. Insufficient venous access for the study procedures.
3. Close affiliation with the investigator, e.g. a close relative of the investigator, dependent person (e.g. employee or student), employee of the department of surgery or nuclear department of the UMCG,TRACER or affiliates.
4. Any finding in the medical examinations or medical history giving, in the opinion of the investigator, reasonable suspicion of a disease or condition that makes treatment with the investigational drug unadvisable, or that might affect interpretation of the results of the study or render the patient at high risk for treatment complications.
5. Participation in an interventional clinical study within 30 days prior to tracer administration that involved treatment with any drug (excluding vitamins and minerals) or medical device.

Medical Exclusion Criteria:

1. The existence of a second concomitant active malignancy or treatment for a second malignancy within 1 year prior to IMP-administration that is not a solid tumor indication included in the VARTUTRACE study, except for localized basal or squamous cell cancer that has been cured at least 90 days before screening.
2. Cardiac impairment with an estimated LVEF <35 % Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the investigator.
3. Any abnormalities in the vital signs of the patient, as judged by the investigator, as a result of which the patient cannot participate. Note: One retest of vital functions is allowed within the screening window.
4. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
5. Major surgical procedure other than for the included diagnosis within four weeks before IMP administration. Disease-related procedures, e.g. the placement of a port-a-cath, placement of a drain, ERCP, are allowed.
6. Current evidence or history of bacterial, viral or fungal infections within 7 days before 89Zr-DFON-Suc-scFv (F8 or C9) administration as judged by the Investigator.

   * T > 38.0°C or lab confirmed viral/bacterial/fungal infection (PCR) or symptoms suggestive of an infection)
   * Received oral or IV antibiotics within <7 days before administration.
7. Any planned major surgery within the duration of the study (until follow-up visit) that is not related to the tumor, with the exception of any emergency surgeries.
8. Prior allogeneic bone marrow transplantation or solid organ transplant.
9. A history of anaphylaxis, history of allergic reaction(s), known allergy to one of the drugs or excipients administered as part of this study. Mild allergies without angio-edema or treatment need can be acceptable if deemed not of clinical significance (including allergy to animals or mild seasonal hay fever).
10. Any other diseases, metabolic dysfunction, physical examination finding, or clinically significant laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Biodistribution and pharmacokinetics of the radiolabeled IMP | Day 1, 2, and 4 after dosing
  Biodistribution and pharmacokinetics of the IMP are defined by the amount of IMP that is taken up per target organ or tissue over time. The radioactive dose absorbed per target organ or tissue over time is determined using whole-body PET/CT imaging at various time points post-injection. In addition, blood samples will be taken at various time points post-injection to determine IMP plasma level concentrations. The ICRP 89 values will be used to calculate the effective dose in each organ. Descriptive statistics of absorbed doses to target organs and tissues specified will be tabulated. The blood concentrations will be presented using descriptive summary statistics.
Tumor-specific uptake of the IMP | Day 1 - 7 after dosing
  Tumor-specific uptake of the IMP is defined as the amount of IMP that tumors uptake compared to normal tissue. Tumor-specific uptake of the IMP is captured using PET/CT imaging and quantified by calculating the tumor-to-background ratio (TBR), which is determined by the ratio of radioactivity taken up by the tumor and radioactivity taken up by healthy reference tissue. A qualified PET investigator will obtain the raw data. PET/CT-derived TBR will be quantified for each patient and compared to standard of care imaging techniques. Variables will be presented as qualitative data. Data interpretation is considered descriptive.
Incidence of treatment emergent adverse events (AE) (safety and tolerability) | Study duration (up to 56 days)
  Safety and tolerability will be assessed by the number of participants with treatment-emergent AEs, with abnormal laboratory tests results (including the occurrence of anti-drug antibodies), abnormal vital signs, abnormal ECG readings, and abnormal physical examination findings from the time of i.v. administration of the IMP until the end of the follow-up period. For this objective, variables will be presented as qualitative data. Interpretations of this data will be descriptive

SECONDARY OUTCOMES:
Tumor-specific uptake of the IMP per cancer type | Day 1 -7 after dosing
  Tumor-specific uptake of the IMP will be quantified, as described in outcome measure 2, for each cancer type and compared across cancer types included in this study. Variables will be presented as qualitative data. Data interpretation is considered descriptive.

OTHER OUTCOMES:
Presence of IMP and target in patient-derived tumor tissue | Day 1 - 7 after dosing
  The presence of the IMP and the oncofetal CS target in tumor tissue will be determined ex vivo and compared to the tracer signal measured in the tumor tissue in vivo. Presence of the IMP and the oncofetal CS target in patient-derived tissue slices will be determined using immunohistochemical stainings. Tumor-specific uptake of the IMP in vivo will be quantified using PET/CT imaging as described in outcome measure 2. For this objective, variables will be presented as qualitative data. Interpretations of this data will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Gooitzen van Dam, MD, PhD, Principal Investigator — TRACER Europe B.V.
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No